CLINICAL TRIAL: NCT01815099
Title: Transcranial Magnetic Stimulation Treatment for Generalized Anxiety Disorder: Substudy #2
Brief Title: Transcranial Magnetic Stimulation Treatment for Generalized Anxiety Disorder
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The remaining eligible participants declined to participate.
Sponsor: Hartford Hospital (Other)
Collaborators: Neuronetics (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DIEF003523.3
Record Dates: First submitted 2012-09-04; First posted 2013-03-20 (Estimated); Results first posted 2017-04-10 (Actual); Last update posted 2017-04-10 (Actual); Status verified 2017-02

CONDITIONS: Generalized Anxiety Disorder
MeSH Terms: conditions — Generalized Anxiety Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- rTMS Treatment (Experimental): Clinical participants will receive rTMS
  Interventions: Device: rTMS Treatment

INTERVENTIONS:
Device: rTMS Treatment — Either 10 or 15 rTMS sessions (2 or 3 times/week for 5 weeks, respectively)
  Other Names: Neurostar

SUMMARY:
We are investigating the feasibility and efficacy of transcranial magnetic stimulation (TMS) for patients with GAD who were placebo nonresponders in DIEF003523.1.

DETAILED DESCRIPTION:
We expected to enroll five patients with GAD who failed to respond to a sham (placebo) TMS intervention. In this pilot study we enrolled three participants into a protocol including 10 rTMS sessions (twice a week for five weeks) and one into a protocol including 15 rTMS sessions (three times a week for five weeks). Assessments occurred at pretreatment and at posttreatment.

ELIGIBILITY:
Inclusion Criteria:

* Participated in the study DIEF003523.1, received sham "placebo" TMS and achieved < 50% improvement in HARS at 3 month follow-up.
* Fluency in English
* Capacity to understand the nature of the study and willingness to sign informed consent form

Exclusion Criteria:

* History of epilepsy or head trauma (LOC > 5 minutes) within the past 6 months
* Lifetime history of increased intracranial pressure, seizure disorder, stroke, brain tumor, multiple sclerosis, or brain surgery
* A review of patient medications by the study physician indicates an increased risk of seizure
* An active autoimmune, endocrine, viral, or vascular disorder affecting the brain; any unstable cardiac disease; hypertension; or severe renal or liver insufficiency
* Substance use disorder or PTSD within the past 6 months
* Lifetime bipolar disorder, obsessive-compulsive disorder (OCD), psychotic disorder, mental retardation, or pervasive developmental disorder
* Any psychotic features, including dementia or delirium
* Concurrent psychotherapy and unwillingness to discontinue
* Medication change within the past 4 weeks
* Current serious suicidal or homicidal ideation, and/or serious suicidal attempt within the past 6 months
* Serious, unstable, or terminal medical condition or clinically judged too psychiatrically unstable to participate in the study
* Any contraindication for participation in MRI scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-05; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gretchen J Diefenbach, Ph.D., Principal Investigator — Hartford Hospital
Locations (1):
- Hartford Hospital, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- rTMS Treatment: This was an open trial. All participants received active rTMS
Period: Overall Study
Arm/Group | rTMS Treatment
Started | 4
Began rTMS Treatment | 3
Completed (For completers: one completed a protocol of 10 sessions and one completed a protocol of 15 sessions) | 2
Not Completed | 2
Not completed — Lack of Efficacy | 1
Not completed — unable to attend study visits | 1

BASELINE CHARACTERISTICS:
Groups:
- rTMS Treatment: rTMS Treatment: will entail twice weekly rTMS sessions for 5 weeks.
Arm/Group | rTMS Treatment
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.75 (15.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in The Structured Interview Guide for the Hamilton Anxiety Rating Scale (SIGH-A) Before and After TMS Treatment.
Description: The Hamilton Anxiety Rating Scale (HARS) is one of the most commonly used and extensively validated outcome measures for anxiety symptoms. The SIGH-A allows for a standardized administration of the HARS. The total score was used in this study. The total score ranges from 0 to 56 with higher scores indicative of more severe anxiety symptoms.
Time Frame: Approximately 1 week prior to initial TMS treatment session, 1 week after final TMS treatment session
Population: rTMS treatment completers
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Pre rTMS Treatment: Assessment before beginning rTMS treatment
- Post rTMS Treatment: Assessment After Completing rTMS
Arm/Group | Pre rTMS Treatment | Post rTMS Treatment
Number analyzed (Participants) | 2 | 2
units on a scale | 20.00 (4.24) | 10.50 (0.71)

ADVERSE EVENTS:
Time Frame: AE data were collected over 5 weeks of treatment
Arm/Group | rTMS Treatment
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | rTMS Treatment (N=3)
pin prick sensation at treatment site (Skin and subcutaneous tissue disorders) | 2
pain or discomfort at treatment site (Skin and subcutaneous tissue disorders) | 3
headache (Nervous system disorders) | 2
eye pain (Eye disorders) | 1
toothache (Musculoskeletal and connective tissue disorders) | 2
face pain (Musculoskeletal and connective tissue disorders) | 2
eye or jaw twitch (Musculoskeletal and connective tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes